CLINICAL TRIAL: NCT00004466
Title: Pilot Study of Atorvastatin in Children With Chronic Hyperlipidemia Secondary to Nephrotic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very poor enrollment
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Southwest Pediatric Nephrology Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199/13924; R21DK053611 (NIH); PD-981-183 (Other: Southwest Pediatric Nephrology Study Group); SPNSG-97.024 (Other: Southwest Pediatric Nephrology Study Group)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Nephrotic Syndrome; Hyperlipidemia
Keywords: cardiovascular and respiratory diseases; hyperlipidemia; nephrotic syndrome; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Nephrotic Syndrome; Hyperlipidemias; Respiratory Tract Diseases; Rare Diseases; Urogenital Diseases | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin
  Arms: Atorvastatin
Drug: Placebo
  Arms: Placebo

SUMMARY:
OBJECTIVES:

I. Determine the effect of atorvastatin on the plasma levels of lipids, Lp(a), and apoproteins for treating hyperlipidemia in children with nephrotic syndrome in whom proteinuria and hyperlipidemia persist after other appropriate measures to treat their primary disease have been exhausted.

II. Determine the safety and tolerability of atorvastatin in these patients.

III. Provide preliminary data for a future investigation into the potential effect that lowering cholesterol levels may have on the rate of progression of renal insufficiency in such patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double blind, placebo controlled, multicenter study.

After 3 months of low cholesterol diet, patients are randomized to receive atorvastatin tablets daily (arm I) or placebo tablets daily (arm II) for 3 months. Arm I patients receive increasing doses of atorvastatin every 4 weeks until individual maximum tolerated doses (MTDs) are determined.

After 3 months of treatment, all patients are given atorvastatin in a 6-9 month open label extended evaluation. Arm I patients receive atorvastatin for an additional 6 months and arm II patients receive atorvastatin for 9 months with increasing doses of atorvastatin every 4 weeks for the first 3 months until MTDs are determined.

Patients are followed every 6-8 weeks for one year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Chronic hyperlipidemia with treatment-resistant nephrotic syndrome; Must have received at least 2 months of therapy with steroids on a daily or alternate basis

Primary nephropathy described as minimal change nephrotic syndrome, mesangioproliferative glomerulonephritis, IgM neuropathy, and focal segmental glomerulosclerosis

Glomerular filtration rate at least 30 mL/min

LDL cholesterol at least 160 mg/dL

--Prior/Concurrent Therapy--

No concurrent medications affecting or interacting with lipids or atorvastatin, with the exception of angiotensin converting enzyme inhibitors at discretion of referring physician, including: lipid-lowering medications, beta blockers, thiazides, fish oils, cyclosporine, Cytoxan, azathioprine, chlorambucil, and erythromycin

Concurrent prednisone and other corticosteroids allowed on a continual basis at a dose of no greater than 1 mg/kg every other day (maximum dose, no greater than 40 mg every other day); Concurrent acute courses of steroids no greater than 1 week for other unrelated conditions (e.g., asthma) also allowed

--Patient Characteristics--

Hepatic: ALT or AST less than 2 times normal

Renal: See Disease Characteristics; Creatine phosphokinase less than 3 times normal

Other: No history of familial hypercholesterolemia; No systemic disease such as systemic lupus, Schoenlein-Henoch purpura, Hodgkin's disease, polyarteritis nodosum, sickle cell disease, or HIV; Not pregnant; Effective contraception required of all adolescent patients

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 1998-10 (Actual); Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma lipid levels | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hogg, Study Chair — Southwest Pediatric Nephrology Study Group
Locations (1):
- Medical City Dallas Hospital, Dallas, Texas, United States